CLINICAL TRIAL: NCT04706026
Title: A Pilot Study of Local Anesthesia for Inguinal Hernia Surgery in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH); American Federation for Aging Research (Other); The John A. Hartford Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0980; Protocol Version 6/26/25 (Other: UW Madison); SMPH/SURGERY/ENDOCRINE (Other: UW Madison); K76AG068515 (NIH); 2025-1446 (Other: UW Madison - UW Health site)
Record Dates: First submitted 2020-12-10; First posted 2021-01-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Inguinal Hernia; Anesthesia, Local
Keywords: Elderly; Outcome; Inguinal hernia; Local anesthesia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: There will be three study arms, participants will be randomized to
  1. Open and laparoscopic / robotic inguinal hernia repair under general anesthesia (Control Group)
  2. Inguinal hernia repair with local anesthesia (Experimental Group)
  An Observational standard of care arm will supplement accrual in each arm to help reach the goal of 80 participants.
Who Masked: Investigator
Masking Description: The investigative team (except for the statistician and the surgeon) will be blinded to the treatment assignment until the final analysis is complete. The study team will not be blinded to the treatment assignments for participants in the observational arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open Inguinal Repair- Local anesthesia (Experimental): This arm will receive local anesthesia for their open inguinal hernia repair.
  Interventions: Other: Open Inguinal Hernia Repair - Local Anesthesia
- Inguinal Hernia Repair- General Anesthesia (Active Comparator): This arm will receive general anesthesia for their open inguinal hernia repair or laparoscopic / robotic repair.
  Interventions: Other: Inguinal Hernia Repair - General Anesthesia
- Observational: Standard of Care (No Intervention): Participants will receive anesthesia and surgery as decided by their care team.

INTERVENTIONS:
Other: Open Inguinal Hernia Repair - Local Anesthesia — Patients in the local anesthesia arm will receive an injection of a 50:50 mix of 1% lidocaine with epinephrine and 0.25% Marcaine at the surgical site (in the skin and subcutaneous layers + beneath the external oblique aponeurosis). Patients in the local arm will also receive intravenous sedation (Propofol or Precedex) and pain medication (morphine or fentanyl) at the discretion of the attending anesthesiologist.
  Arms: Open Inguinal Repair- Local anesthesia
Other: Inguinal Hernia Repair - General Anesthesia — General anesthesia will be administered at the discretion of the anesthesiologist and will involve a combination of inhaled and intravenous anesthesia.
  Arms: Inguinal Hernia Repair- General Anesthesia

SUMMARY:
The purpose of this study is to collect data about local versus general anesthesia for inguinal hernia repair in Veterans aged 60 years for planning a larger, multisite randomized clinical trial. Approximately 80 participants will be enrolled and can expect to be on study for 6 months.

DETAILED DESCRIPTION:
The study rationale is that prior to conducting a multisite randomized trial, it is necessary to identify relevant outcomes, understand barriers to greater use of local anesthesia, test study procedures, and confirm our ability to adequately recruit and randomly assign participants. Additionally, the proposed study will provide the applicant with critical training in the design, conduct, and analysis of clinical trials. This will uniquely position the applicant to change surgical care for older adults.

More specifically, the investigators plan to demonstrate the ability to successfully randomize Veterans aged 60 years and older to local versus general anesthesia for inguinal hernia surgery, and to validate processes and instruments to measure relevant outcomes.

Although the original NIA-approved proposal involved only two arms, open hernia repair using local anesthesia and open repair using local anesthesia, the study team subsequently published a paper that showed using local anesthesia for open hernia repair may also be superior to laparoscopic or robotic hernia repair. Consequently, a third arm is added to our pilot study: laparoscopic or robotic hernia repair with general anesthesia (these surgical approaches cannot be done using local anesthesia). The rationale is that use of laparoscopic or robotic inguinal hernia surgery, while still less common than open repair, is becoming more common and no prior randomized trials have compared laparoscopic/robotic surgery versus open repair using local anesthesia.

Local or general anesthesia are the primary methods of anesthesia for inguinal hernia surgery for most surgeons (though some perform the operation under spinal or regional anesthesia, this is rare). Both approaches are used in clinical practice with acceptable known risks and complications. General anesthesia is associated with risks of hypotension, venous thromboembolism, heart attack, stroke, pulmonary dysfunction, cognitive dysfunction, allergic reaction, urinary retention, and malignant hyperthermia. The main risks of local anesthesia include allergic reaction and hypotension (when the anesthetic is improperly injected into a blood vessel).

The primary objective is to:

1. demonstrate ability to successfully recruit, randomize, and retain patients aged 60 years and older for a randomized trial of local versus general anesthesia for inguinal hernia surgery, and
2. establish the ability to measure relevant outcomes and test protocols and study instruments for measuring key outcomes.

The secondary objective is to generate preliminary comparisons between the study arms, to inform effect size estimates for a larger multisite trial.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 60 years
* Presenting to clinic with a unilateral inguinal hernia that is not incarcerated
* Considered suitable for either general or local anesthesia
* Willing to complete all study requirements, including follow-up continuing until six months after surgery
* English speaking

Exclusion Criteria:

* The hernia that the patient is being evaluated for has undergone prior repair
* Any contraindications to general anesthesia
* Allergies to local anesthesia
* Evidence of hernia incarceration or strangulation
* Active local or systemic infection that would preclude the use of mesh for hernia repair
* Need for concurrent surgical repair at the time of hernia repair
* English is not the patient's primary language
* Enrollment in other research studies
* Clinical judgement of surgeon or anesthesiology
* Current pregnancy
* Unwilling to provide consent
* Current active illegal drug use
* Current alcoholism
* Claustrophobia
* Unable to tolerate lying in supine position for greater than 30 minutes

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Rates of enrollment and percentage of eligible patients enrolled | Through study completion, estimated 2 years
  Each week, research assistants will compile running counts of patients screened, found eligible, and enrolled.
Proportion of participants completing all study visits | Through study completion, estimated 2 years
  Assistants will maintain counts of participants who complete each study visit.
Proportion of missing data | Through study completion, estimated 2 years
  At each visit, every study visit will be entered into our electronic database and missing items will have a separate code number.
Time to complete study evaluations and instruments | Time from beginning to end of completing study instrument, up to 2 hours
  Assistants will time participants while completing each study research form and will time the entire encounter.
Participant satisfaction | At 6 month follow up
  A 10 point likert scale will measure participant satisfaction. Scores range from 1-10 with higher scores indicating higher satisfaction.
Whether Survey Instruments Can Be Eliminated due to Redundancy measured by R2 greater than 40% | measured at 25 percent of planned enrollment and 75 percent of planned enrollment, estimated to be up to 1.5 years
  Each survey instrument will be evaluated as the dependent variable in a separate linear regression with the scores of all other instruments used as predictors, along with demographic information. The adjusted R2 (explained variance) for each regression will be estimated. Any instrument where the R2 exceeds 40% will be eliminated based on the idea that little additional information is provided by including that instrument (i.e., the other surveys explain a substantial portion of the information contained within that instrument).
Estimate sample size for fully powered randomized trial | Final sample size estimate will be performed after data collection for the last patient is complete, estimated up to 2 years
  For continuous variables, means and standard deviations will be estimated. For categorical variables, estimated proportions and 95% confidence intervals.

SECONDARY OUTCOMES:
Carolinas Comfort Scale Score | Measured at baseline, 48 hours after surgery, 2 weeks after surgery, 6 months after surgery
  The Carolinas Comfort Scale measures quality of life. Possible scores range from 1-6 for each item, with higher scores indicating increased quality of life.
Physical Function Score | Measured at baseline, 48 hours after surgery, 2 weeks after surgery, 6 months after surgery
  The patients' ability to perform their activities of daily living will be measured with the 6 item Katz index. This scale is from 0-6, with higher scores indicating more functional independence.
Trail Making Test | Measured at baseline, prior to discharge, 48 hours after discharge, 2 weeks after surgery, 6 months after surgery
  Trail Making Test will be used to measure cognitive function. The time to complete the trail making test is measured, with those taking greater than expected time being considered deficient.
Montreal Cognitive Assessment | Measured at baseline, prior to discharge, 48 hours after discharge, 2 weeks after surgery, 6 months after surgery
  Montreal Cognitive Assessment 5 minute form to measure cognitive function. For the Montreal Cognitive Assessment, the successfully completed skills are added to achieve a final score from 0-30, with higher numbers indicating closer to normal cognitive function.
Participants with Delirium | Measured at baseline, prior to discharge, 48 hours after discharge, 2 weeks after surgery, 6 months after surgery
  The Confusion Assessment Method short form consists of 5 questions, if inattention + acute onset and/or fluctuating course + Disorganized thinking and/or Altered level of consciousness are present this test is considered positive for delirium.
Pain Level | Measured at baseline, prior to discharge, 48 hours after discharge, 2 weeks after surgery, 6 months after surgery
  10 point visual analog scale. Patients indicate on a scale of 0-10 their current level of pain. Higher numbers indicate higher pain.
Postoperative complications | Up to 2 weeks
  All complications will be recorded based on VA Surgical Quality Improvement Program definitions.
Operative time | Time between surgery start and surgery end measured. 1 day of surgery
  The amount of time the surgery takes (minutes)
Anesthesia time | Time spent in operating room. 1 day of surgery
  The amount of time in the operating room (minutes)
Recovery time | Time spent in post anesthesia care unit. 1 day of surgery
  Time spent in the post anesthesia care unit and stepdown units.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Balentine, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No